CLINICAL TRIAL: NCT03701932
Title: Mental Activity During Transcranial Magnetic Stimulation (TMS) Therapy for Depression
Brief Title: Mental Activity During (TMS) Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Lumos Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Peter Rosenquist, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 663245
Record Dates: First submitted 2018-03-26; First posted 2018-10-10 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Impairment
Keywords: Depression, Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS and Lumosity® cognitive retraining (Experimental): Group will receive TMS and will concurrently engage in cognitive retraining exercises comprised of the Lumosity® battery.
  Interventions: Behavioral: TMS and Lumosity®cognitive retraining
- TMS and non cognitive computer games (Active Comparator): Group will receive TMS while concurrently engaging in selected computer games from several gaming software that includes Play 101 Games and Hoyle Puzzle and Board Games®. They will also be allowed to spend time on gaming activities of their choice in order to keep them engaged
  Interventions: Behavioral: TMS and non cognitive computer games

INTERVENTIONS:
Behavioral: TMS and Lumosity®cognitive retraining — The Lumosity® training includes exercises for speed, memory, attention, flexibility, and problem solving. Subjects will complete this battery while receiving TMS treatment.
  Arms: TMS and Lumosity® cognitive retraining
Behavioral: TMS and non cognitive computer games — Subjects will play computer games while receiving TMS treatment.
  Arms: TMS and non cognitive computer games

SUMMARY:
The purpose of the study is to assess the effects of different types of mental activity performed while receiving transcranial magnetic stimulation (TMS) for the treatment of major depressive disorder. Our primary aim for this study is to assess the feasibility of combining TMS and computer based cognitive exercise in patients with major depressive disorder who may also have some degree of cognitive dysfunction, and to formally measure changes in mood and cognition over the course of the study.

DETAILED DESCRIPTION:
Patients will receive TMS treatment daily for 6 weeks as part of their standard care. They will complete clinical assessments and participate in cognitive retraining through completion of 15 hours of Lumosity gaming cognitive exercises while simultaneously receiving active TMS stimulation. Those participants in the control group will complete 15 hours of computer gaming activity during the administration of active stimulation. Computer games in the control group exercises are elected by the patient from a library of intellectually and motivationally engaging games drawn from several gaming software compilations that includes Play 101 Games and Hoyle Puzzle and Board Games.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has a diagnosis of depression

  * Subject has been approved and scheduled to receive TMS at Augusta University
  * Subject does not have a major neurocognitive impairment or an alcohol or substance abuse disorder, and can see images on a computer monitor.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The University of Pennsylvania Computerized Neuropsychological Testing Battery (Penn CNP) | Change from baseline at six weeks
  Administers computerized neuropsychological tests for research studies

SECONDARY OUTCOMES:
The Lumosity® Brain Performance Test (BPT) | Change from baseline at six weeks
  Online neuropsychological battery of assessments measuring training-related changes in Cognitive Performance
Inventory of Depressive Symptoms- Self Report | Change from baseline at six weeks
  Patient rating of depressive symptom severity
Hamilton Depression Rating Scale 17 item | Change from baseline at six weeks
  Clinician Rating of Depressive Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Rosenquist, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No